CLINICAL TRIAL: NCT01069783
Title: A Phase IIa, Double-blind, Randomised, Placebo-controlled, Dose-finding Efficacy and Safety Study of A3309 in Patients With Dyslipidemia
Brief Title: Study of A3309 in Patients With Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3309-005
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Dyslipidemia
Keywords: dyslipidemia; cholesterol; LDL
MeSH Terms: conditions — Dyslipidemias | interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A3309 low dose (Experimental)
  Interventions: Drug: A3309
- A3309 high dose (Experimental)
  Interventions: Drug: A3309
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: A3309 — A3309 in two different dosage levels
  Arms: A3309 high dose; A3309 low dose
Drug: A3309 — A3309 in two different dosage levels for the duration of the study
  Arms: A3309 high dose; A3309 low dose
Drug: Placebo — Placebo comparator once daily for the duration of the trial
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of A3309 administered to patients with dyslipidemia (high cholesterol levels).

ELIGIBILITY:
Inclusion Criteria:

* Patients meet protocol specified criteria for dyslipidemia and has successfully completed study requirements with no clinically relevant findings

Exclusion Criteria:

* Medical history or medical condition that would not make the patient a good candidate for the study or would limit the patient´s capability to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low-density lipoprotein (LDL) cholesterol | eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- BCRC, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants. Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Rudling M, Camilleri M, Graffner H, Holst JJ, Rikner L. Specific inhibition of bile acid transport alters plasma lipids and GLP-1. BMC Cardiovasc Disord. 2015 Jul 22;15:75. doi: 10.1186/s12872-015-0070-9. PMID 26197999